CLINICAL TRIAL: NCT01418898
Title: The Effect of a Nutrient Fortified Oat Drink on Iron, Zinc, Vitamin A, and Vitamin C Status Among Filipino Children
Brief Title: Nutrient Fortified Oat Drink
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PepsiCo Global R&D (Industry)
Collaborators: PepsiCo - Philippines (Unknown)
Responsible Party: Imelda Angeles-Agdeppa, Ph.D, Food and Nutrition Research Institute Department of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PEP 1011
Record Dates: First submitted 2011-08-15; First posted 2011-08-17 (Estimated); Last update posted 2011-08-17 (Estimated); Status verified 2011-08

CONDITIONS: Iron Deficiency Anemia
Keywords: Iron deficiency anemia; iron; zinc; vitamin A; vitamin C; oats
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutrient Fortified Beverage (Experimental)
  Interventions: Other: Dietary Intervention
- Control (Placebo Comparator)
  Interventions: Other: Dietary Intervention

INTERVENTIONS:
Other: Dietary Intervention — Nutrient fortified oat beverage

SUMMARY:
This study will follow a randomized, double-blind, placebo-controlled, parallel-group design to test if an oat beverage fortified with iron, zinc vitamin A and vitamin C will improve nutrient status and iron deficiency in young children compared to an unfortified control beverage.

ELIGIBILITY:
Inclusion Criteria:

* 5-7 years old
* Children with parental consent
* Not suffering from diarrhea, respiratory infections and fever at time of interview and for the past two weeks
* No history of blood disorder or malaria
* Had not participated in any feeding program for the past 4 months
* Children with Hb > 70 g/L to <120 g/L (WHO/UNICEF/UNU, 1998)
* CRP <10 mg/L

Exclusion Criteria:

* All children aged < 5 years old and > 7 years old
* Without parental consent
* Undergoing treatment for any chronic ailment, diagnosed as suffering from any sort of illness e.g. fever, diarrhea, stomach ache, cough and colds at the time of examination or during the past two weeks.
* Reported current or history of blood abnormalities/hemoglobinopathies
* Children with all normal Hb levels or very low Hb < 70 g/L
* CRP >10mg/L

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2011-08; Primary Completion 2011-12 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Iron status: Change in hemoglobin and serum ferritin | Baseline and 4 months

SECONDARY OUTCOMES:
zinc, vitamin A and vitamin C status | Baseline and 4 months
Weight, height, CRP and frequency of illness | Baseline and 4 months
Dietary intake | Baseline and 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Imelda Angeles-Agdeppa, PhD, Principal Investigator — FNRI
Locations (1):
- FNRI, City of Taguig, Philippines